CLINICAL TRIAL: NCT05851807
Title: Intraoperative Lung Mechanics, Postoperative Complications, and Functional Evaluation in Post COVID-19 Patients Undergoing Thoracic Surgery
Brief Title: Intraoperative Lung Mechanics and Functional Evaluation in Post COVID-19 Thoracotomy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Associated Professor Dr, Ankara University
Other Study IDs: i04-208-22
Record Dates: First submitted 2023-05-08; First posted 2023-05-10 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pandemic; Anesthesia; Thoracic Diseases
Keywords: Covid-19; Thoracic Anesthesia
MeSH Terms: conditions — COVID-19; Thoracic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patints with COVID-19 History: Patients with infected with COVID-19 in any time.
- Patints without COVID-19 History: Patients without COVID-19 history.

SUMMARY:
At the end of 2019, cases of an unknown respiratory infection were reported in the city of Wuhan in China. It was determined that the cause of this infection was a new virus belonging to the coronavirus family, which was named SARS-CoV-2. After the virus spread worldwide, the World Health Organization (WHO) declared it a pandemic. The clinical picture and disease caused by the virus were named COVID-19 (1). According to the WHO's data on 29.01.2022, the number of cases worldwide has exceeded 365 million, and the number of deaths has exceeded 5 million (2). Fever, cough, fatigue, shortness of breath, myalgia, sore throat, and headache are the main symptoms of COVID-19. Less frequently, it can cause nausea, vomiting, and diarrhea. The disease has a broad spectrum ranging from mild illness to severe illness that can result in death (3). In a study analyzing the data of approximately 72,000 patients in China, it was reported that 81% of the patients had no lung involvement or minimal involvement, 14% had severe involvement, and 5% had respiratory failure, shock, or multiple organ failure (4).

Attention is drawn to the long-term complications of COVID-19, such as myocarditis, heart failure, arrhythmia, dyspnea, oxygen dependence, impaired respiratory function tests, increased venous/arterial thromboembolism, decreased fitness, muscle and joint pain, increased anxiety-depression, post-traumatic stress disorder, and renal damage (5). It has been emphasized that patients who have recovered from COVID-19, especially older individuals and those with severe illness, are at risk of sarcopenia (7). It has been suggested that in patients who have recovered from COVID-19, direct viral damage, decreased physical activity level, and malnutrition result in decreased fitness and sarcopenia, which could be associated with increased morbidity in cancer surgeries (8).

It is reported that postoperative complications and deaths are higher in active COVID-19 patients than in those who do not have active disease (9). In a multicenter study, it was stated that postoperative pulmonary complications were observed in half of the patients who had COVID-19 during the perioperative period, and this condition was associated with high mortality. Most of these patients are those who need emergency surgical interventions (10).

According to studies in the literature, COVID-19 has multi-systemic effects, and some of these effects continue in the long term. It has been shown that the perioperative period with COVID-19 positivity is associated with higher pulmonary complications and mortality. It has been suggested that having had COVID-19 in the past may lead to worse postoperative outcomes. The studies in the literature were mostly conducted on patients who had surgery during the perioperative period while having COVID-19. Most of the patients required emergency surgical interventions. The effect of the patients' functional level on postoperative outcomes has not been examined. Our study focuses on the intraoperative and postoperative period of thoracic surgery patients who underwent surgery in the long term after COVID-19.

DETAILED DESCRIPTION:
Patients over the age of 18, who are planned to undergo thoracotomy, will be recruited. Those volunteers whose COVID-19 infection is confirmed by PCR test will form the COVID-19 patient group, while others will form the control group who did not have COVID-19. The patient group to be operated on and followed by the Department of Thoracic Surgery of the Ankara University, Faculty of Medicine will be analyzed.

Before starting the evaluations, the patients will be asked to review the informed consent form and give their consent to participate in the research. The sociodemographic data (name, surname, file number, date of birth, height, weight, marital status, education level, occupation, contact number) and medical history (systemic diseases and their duration, drugs used continuously and their duration) of the patients who agree to participate in the study will be recorded.

The ASA (American Society of Anesthesiologists) score will be determined in the preoperative period. Hemoglobin values before the operation will be recorded. It will be queried whether the participants had COVID-19, and in the group that had it, the date of COVID-19 infection, whether oxygen therapy was received before COVID-19, inhaler and BPAP-CPAP usage status, the presence of COPD, severe emphysema, uncontrolled asthma, OSAS (Obstructive sleep apnea syndrome), or previous pulmonary surgery history will be recorded. It will be queried whether imaging was performed with computed tomography during COVID-19 diagnosis and follow-up, and if performed, whether there was lung involvement and its percentage will be recorded. Medical treatments received by the patient during COVID-19, need for ventilation support will be noted. The duration of hospitalization in the inpatient and intensive care units due to COVID-19 will be recorded. The need for oxygen support after discharge due to COVID-19 will be queried. ARISCAT scores will be determined in both groups. Arterial blood gas results taken before the operation will be recorded. Predicted postoperative forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), and DLCO (diffusing capacity of the lung for carbon monoxide) values will be determined before the operation.

Jamar dynamometer will be used to measure grip strength (Mathiowetz 1984). Assessment with Jamar dynamometer will be performed during the preoperative assessment, discharge phase, and 1-month control after the operation. Patients will be asked to squeeze the dynamometer as hard as they can while their upper extremities are positioned appropriately. Measurements will be taken three times for each side.

To evaluate lower extremity muscle strength and balance, a 5-repetition sit-to-stand test will be applied (Munoz-Bermejo 2021). This test will be performed during the preoperative assessment, discharge phase, and 1-month control after the operation. Patients will be asked to stand up from the chair five times while sitting on the chair. The time required for each patient to complete the test will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* The Informed Consent Form must be signed by the patient
* Being over 18 years old
* The plan is to undergo pneumonectomy, lobectomy, segmentectomy, or various degrees of lung resection surgery

Exclusion Criteria:

* Informed Voluntary Consent Form not signed by the patient
* The presence of contraindications for the administration of cardiopulmonary exercise testing
* Lack of mental and psychological competence to complete the assessment and testing phases The presence of musculoskeletal problems that could hinder the implementation of evaluation and testing stages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There has not been a similar study before, and in this respect, the study is a pilot study. Considering the number of patients who underwent lung resection and required evaluation with CPET in the Department of Thoracic Surgery of Ankara University Faculty of Medicine, the average annual number of operations is 250, and the number of patients for 3 years is predicted to be 750 in total. Considering the inclusion and exclusion criteria of the study, the number of patients was determined as 60 patients in the COVID-19 group and 60 patients in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-05-12 (Estimated); Study Completion 2024-05-12 (Estimated)

PRIMARY OUTCOMES:
significant difference in cardiopulmonary exercise capacity during and after thoracic surgery | 1 month
  There is a significant difference in cardiopulmonary exercise capacity during and after thoracic surgery between patients who have had COVID-19 and those who have not.

SECONDARY OUTCOMES:
significant difference in muscle strenght | 1 month
  There is a significant decrease in the 6-minute walking distance and grip strength after thoracic surgery in patients who have had COVID-19 compared to those who have not. Additionally, there is a significant increase in the duration of the 5-repetition sit-to-stand test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atzrodt CL, Maknojia I, McCarthy RDP, Oldfield TM, Po J, Ta KTL, Stepp HE, Clements TP. A Guide to COVID-19: a global pandemic caused by the novel coronavirus SARS-CoV-2. FEBS J. 2020 Sep;287(17):3633-3650. doi: 10.1111/febs.15375. Epub 2020 Jun 16. PMID 32446285
- [Background] Chams N, Chams S, Badran R, Shams A, Araji A, Raad M, Mukhopadhyay S, Stroberg E, Duval EJ, Barton LM, Hajj Hussein I. COVID-19: A Multidisciplinary Review. Front Public Health. 2020 Jul 29;8:383. doi: 10.3389/fpubh.2020.00383. eCollection 2020. PMID 32850602
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Desai AD, Lavelle M, Boursiquot BC, Wan EY. Long-term complications of COVID-19. Am J Physiol Cell Physiol. 2022 Jan 1;322(1):C1-C11. doi: 10.1152/ajpcell.00375.2021. Epub 2021 Nov 24. PMID 34817268
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Welch C, Greig C, Masud T, Wilson D, Jackson TA. COVID-19 and Acute Sarcopenia. Aging Dis. 2020 Dec 1;11(6):1345-1351. doi: 10.14336/AD.2020.1014. eCollection 2020 Dec. PMID 33269092
- [Background] Casey P, Ang Y, Sultan J. COVID-19-induced sarcopenia and physical deconditioning may require reassessment of surgical risk for patients with cancer. World J Surg Oncol. 2021 Jan 11;19(1):8. doi: 10.1186/s12957-020-02117-x. PMID 33430881
- [Background] Doglietto F, Vezzoli M, Gheza F, Lussardi GL, Domenicucci M, Vecchiarelli L, Zanin L, Saraceno G, Signorini L, Panciani PP, Castelli F, Maroldi R, Rasulo FA, Benvenuti MR, Portolani N, Bonardelli S, Milano G, Casiraghi A, Calza S, Fontanella MM. Factors Associated With Surgical Mortality and Complications Among Patients With and Without Coronavirus Disease 2019 (COVID-19) in Italy. JAMA Surg. 2020 Aug 1;155(8):691-702. doi: 10.1001/jamasurg.2020.2713. PMID 32530453
- [Background] COVIDSurg Collaborative. Mortality and pulmonary complications in patients undergoing surgery with perioperative SARS-CoV-2 infection: an international cohort study. Lancet. 2020 Jul 4;396(10243):27-38. doi: 10.1016/S0140-6736(20)31182-X. Epub 2020 May 29. PMID 32479829
- [Background] Mathiowetz V, Weber K, Volland G, Kashman N. Reliability and validity of grip and pinch strength evaluations. J Hand Surg Am. 1984 Mar;9(2):222-6. doi: 10.1016/s0363-5023(84)80146-x. PMID 6715829
- [Background] Munoz-Bermejo L, Adsuar JC, Mendoza-Munoz M, Barrios-Fernandez S, Garcia-Gordillo MA, Perez-Gomez J, Carlos-Vivas J. Test-Retest Reliability of Five Times Sit to Stand Test (FTSST) in Adults: A Systematic Review and Meta-Analysis. Biology (Basel). 2021 Jun 9;10(6):510. doi: 10.3390/biology10060510. PMID 34207604
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414
- [Background] Lollgen H, Leyk D. Exercise Testing in Sports Medicine. Dtsch Arztebl Int. 2018 Jun 15;115(24):409-416. doi: 10.3238/arztebl.2018.0409. PMID 29968559
- See also: Related Info — https://covid19.who.int